CLINICAL TRIAL: NCT05793164
Title: Characterization and Risk Factors of Folliculitis After Hair Transplantation
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2020-152
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Folliculitis
Keywords: folliculitis; hair transplantation; Follicular Unit Extraction
MeSH Terms: conditions — Folliculitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with postoperative folliculitis: Patients presented folliculitis in surgical-area lesions after hair transplantation within 9-month follow up.
  Interventions: Other: no intervention
- patients without postoperative folliculitis: Patients didn't present folliculitis in surgical-area lesions after hair transplantation within 9-month follow up.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
We retrospectively reviewed 1317 patients who had undergone HT and completed 9-month follow-up between January 2018 and June 2021 at 4 medical centers. The incidence of postoperative folliculitis and the patient demographics were assessed. Logistic regression analysis was used to identify the risk factors, and the characteristics of different types of folliculitis were compared.

DETAILED DESCRIPTION:
Postoperative folliculitis is a common complication after hair transplantation (HT) and requires effective preventive interventions. This study aimed to characterize postoperative folliculitis and determine the risk factors in patients underwent HT. The study was conducted at 4 clinical sites: Nanfang Hospital of Southern Medical University, the First Affiliated Hospital, Zhejiang University School of Medicine, the Affiliated Hospital of Guilin Medical University, and Peking University Third Hospital. Data of 1317 patients who had undergone HT and completed a 9-month follow-up from January 2018 to June 2021 were collected. The incidence of postoperative folliculitis and the patient demographics were assessed. Logistic regression analysis was used to identify the risk factors, and the characteristics of different types of folliculitis were compared.

ELIGIBILITY:
Inclusion Criteria:

- 1. Healthy adults between the ages of 18 ~ 60

2. patients suitable for autologous hair transplantation according to "the standard of hair transplantation"

Exclusion Criteria:

1. Coagulation disorders, pregnancy and lactation, immunosuppression
2. With severe mental and psychological illness, impairment of body image
3. All kinds of immune-related alopecia in the progressive active stage
4. Patients judged by the investigator to be unsuitable for this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Data of 1317 patients who had undergone HT and completed a 9-month follow-up from January 2018 to June 2021 were collected.
Sampling Method: Probability Sample
Enrollment: 1317 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
folliculitis | 9 months after hair transplantation
  patients present folliculitis after hair transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Zhiqi Hu, PhD, Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China